CLINICAL TRIAL: NCT02636127
Title: Role of Circulating Cytotoxic Lymphocytes in Endothelial Cell Injury in Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015-37
Record Dates: First submitted 2015-12-09; First posted 2015-12-21 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systemic Sclerosis (SSc) patient (Experimental): 15 patients whose diagnosis of SSc is made according to the revised ACR/EULAR ( American College of Rheumatology ) criteria 2013 will be recruited and blood samples will be obtained
  Interventions: Other: blood samples
- healthy patient (Other): 15 healthy patients will be recruited and blood samples will be obtained
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — one blood sample will be done for dosage and role of Fractalkine in the serum.
  - Functional study of the interactions between T cells and NK cells and / endothelial cells (HMVEC): immuno mediated endothelial cytotoxicity, endothelial activation and microparticles release by the HMVEC, endothelial progenitor cells analysis and evaluation of the endothelial lysis by fluorescence release.

SUMMARY:
Systemic Sclerosis (SSc) is an auto-immune systemic disease characterized by vascular damage, cutaneous and visceral fibrosis and a dysimmune condition.

Therapies in this disease remain insufficient and the complications resulting from organs involvement lead to strong morbi-mortality.The dermic infiltrate of the patients includes a strong proportion of Tcells. T cells and Natural Killer (NK) cells are potentially involved in the vascular damage of the SSc. However mechanisms at the onset of this endothelial cytotoxicity and its impact on the capacities of regeneration of the endothelial tissue remain poorly understood. Fractalkine is at the same time an endothelial membrane-bound adhesion molecule and a chemokine which is able to bind CX3CR1 expressed by the immune populations. The purpose of the project is to define the role displayed by cytotoxic, circulating immune populations of SSc patients in endothelial cytotoxicity as well as the role of the axis Fractalkine / CX3CR1 in mediating the interactions between the immune cytotoxic cells and the endothelium.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by SSc of more than 18 years
* Healthy patients

Exclusion Criteria:

* Impossibility to take some blood
* Current infection
* Ongoing cancer
* chemotherapy or a current radiotherapy
* pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2016-07-21 (Actual); Study Completion 2018-07-08 (Actual)

PRIMARY OUTCOMES:
blood sample will be done for dosage of Fractalkine in the serum | 12 months

SECONDARY OUTCOMES:
blood sample for functional study of the interactions between T cells and NK cells and / endothelial cells (HMVEC) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte GRANEL, MD, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No